CLINICAL TRIAL: NCT05169905
Title: A Phase III, Randomized, Open-label, Active Vaccine-controlled Crossover Study to Evaluate the Reactogenicity, Safety and Immune Response of Unadjuvanted RSV Maternal Vaccine in Healthy Non-pregnant Girls From 9 to 17 Years of Age, and in Non-pregnant Adult Women From 18 to 49 Years of Age
Brief Title: A Study to Evaluate the Safety and Immune Response to an Unadjuvanted RSV Maternal Vaccine in Healthy Non-pregnant Females From 9 to 49 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 217354; 2021-004003-41 (EudraCT Number)
Record Dates: First submitted 2021-12-10; First posted 2021-12-27 (Actual); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus Maternal vaccine; Combined reduced-antigen-content diphtheria, tetanus and acellular pertussis vaccine; Reactogenicity; Safety; Immunogenicity; Healthy non-pregnant girl; Healthy non-pregnant adult women
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Tetanus | interventions — Boostrix

STUDY DESIGN:
Intervention Model Description: The interventional study model was planned to be crossover, but this is no longer applicable as there were no more study activities planned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- RSV_dTpa-P Group (Experimental): Healthy non-pregnant girls 9-17 years of age received a single dose of RSV MAT vaccine at Day 1 and were scheduled to receive a single dose of dTpa vaccine at Day 31 and to be followed-up until end of study (180 days post-vaccine administration). Participants who were enrolled and were due to receive the dTpa vaccine at Day 31, did no longer receive the dTpa as part of this study, but they were provided with an option to decide to receive dTpa vaccination as part of standard of care/local recommendation on immunization.
  Interventions: Combination Product: RSV MAT vaccine; Combination Product: dTpa vaccine
- dTpa_RSV-P Group (Experimental): Healthy non-pregnant girls 9-17 years of age were scheduled to receive a single dose of dTpa vaccine at Day 1 and a single dose of RSV MAT vaccine at Day 31 and to be followed-up until end of study (180 days post-vaccine administration), but there were no participants assigned to this study group, and hence, there was no vaccine administered in this study group.
  Interventions: Combination Product: RSV MAT vaccine; Combination Product: dTpa vaccine
- RSV_dTpa-A Group (Experimental): Healthy non-pregnant adult women 18-49 years of age received a single dose of RSV MAT vaccine at Day 1 and were scheduled to receive a single dose of dTpa vaccine at Day 31 and to be followed-up until end of study (180 days post-vaccine administration). Participants who were enrolled and were due to receive the dTpa vaccine at Day 31, did no longer receive the dTpa as part of this study, but they were provided with an option to decide to receive dTpa vaccination as part of standard of care/local recommendation on immunization.
  Interventions: Combination Product: RSV MAT vaccine; Combination Product: dTpa vaccine
- dTpa_RSV-A Group (Experimental): Healthy non-pregnant adult women 18-49 years of age received a single dose of dTpa vaccine at Day 1 and were scheduled to receive a single dose of RSV MAT vaccine at Day 31 and to be followed-up until end of study (180 days post-vaccine administration). RSV MAT vaccine was no longer administered to participants at Day 31.
  Interventions: Combination Product: RSV MAT vaccine; Combination Product: dTpa vaccine

INTERVENTIONS:
Combination Product: RSV MAT vaccine — Single dose of the RSV MAT vaccine reconstituted with NaCl solution was planned to be administered intramuscularly, in the non-dominant arm, at Day 1 or at Day 31, depending on the vaccination schedule.
  RSV MAT vaccine was no longer administered to participants at Day 31. No vaccine was administered in the dTpa_RSV-P Group, since there were no participants assigned to it.
Combination Product: dTpa vaccine — Single dose of the dTpa vaccine was planned to be administered intramuscularly, in the non-dominant arm, at Day 1 or at Day 31, depending on the vaccination schedule.
  Two formulations of dTpa vaccine are licensed in the US and outside of the US (ex-US), respectively. dTpa-US formulation was administered to participants in centers located in the US, while dTpa-ex-US formulation was planned to be administered to participants in centers ex-US. The dTpa-ex-US formulation was not applicable in this study anymore as no non-US sites were initiated before the decision to stop the study.
  The participants in RSV_dTpa-P and RSV_dTpa-A study groups were provided with an option to decide to receive dTpa vaccination as part of standard of care/local recommendation on immunization.
  No vaccine was administered in the dTpa_RSV-P Group, since there were no participants assigned to it.
  Other Names: Boostrix

SUMMARY:
The purpose of this study was to evaluate the reactogenicity, safety and immune response of a single intramuscular dose of the respiratory syncytial virus maternal (RSV MAT) vaccine in healthy non-pregnant girls 9-17 years of age (YOA) compared to non-pregnant adult women 18-49 YOA. The combined reduced-antigen-content diphtheria, tetanus and acellular pertussis (dTpa) vaccine was planned to be used as an active control for safety and reactogenicity evaluation.

Following a recommendation from the Independent Data Monitoring Committee of NCT04605159 (RSV MAT 009), GSK made the decision to stop enrolment and vaccination in this study. Enrolled study participants were monitored as part of the study until study completion.

ELIGIBILITY:
Inclusion Criteria:

Healthy Non-pregnant Adult Women from 18-49 YOA

* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the participant prior to performance of any study-specific procedure.
* A healthy female participant, as established by medical history and clinical examination, between and including 18 to 49 YOA at the time of the first study intervention administration.
* Body mass index (based on participant's report) 17.0 to 39.9 kg/m^2, inclusive for adult participants.
* Female participants of childbearing potential may be enrolled in the study, if the participant:

  * has practiced adequate contraception for 1 month prior to study intervention administration, and
  * has a negative pregnancy test on the day of study intervention administration, and
  * has agreed to continue adequate contraception during the entire treatment period and for 1 month after completion of the study intervention administrations.
* Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.

Healthy non-pregnant Girls from 9-17 YOA

* Participants and participants' parent(s)/Legally Acceptable Representative(s) (LAR), who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the participant*/parent(s)/LAR(s) of the participant prior to performance of any study-specific procedure.

  * *Written informed consent obtained from parents/LARs and written informed assent obtained from the participant if she is less than legal age. The legal age is determined according to local regulations in each participating country.
  * In case the legal age is achieved during the conduct of the study, an additional written informed consent from the participant should be obtained at the time of the legal age.
* A healthy female participant between and including 9 and 17 YOA at the time of the first study intervention administration.

  * Female participants of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, or bilateral ovariectomy.
* Body mass index by age between 5 percentile and 95 percentile (inclusive) for pediatric participants.
* Female participants of childbearing potential may be enrolled in the study, if the participant:

  * has a negative pregnancy test on the day of study intervention administration, and is abstinent during the entire treatment period and for 1 month before and after completion of the study intervention administration series (and if so, this is to be documented in the source documents at each vaccination visit)
  * or has practiced adequate contraception for 1 month prior to study intervention administration and has agreed to continue adequate contraception during the entire treatment period and for 1 month after completion of the study intervention administration series.

Exclusion Criteria:

Medical conditions

* Any clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study intervention(s).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Current autoimmune disorder (based on medical history and physical examination), for which the participant has received immune-modifying therapy within 6 months, before study vaccination.
* Hypersensitivity to latex.
* Acute or chronic clinically significant abnormality or poorly controlled pre-existent co-morbidities or any other clinical conditions, as determined by physical examination or medical history that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
* Significant or uncontrolled psychiatric illness.
* Documented human immunodeficiency virus (HIV)-positive participant.
* Any clinically significant* hematological parameter and/or biochemical laboratory abnormality from the test requested by the investigator based on medical judgment prior to enrolment

  * *The investigator should use his/her clinical judgment to decide whether the test is needed, and which abnormalities are clinically significant. If he/she decides to run this test, the investigator will need to review the test results before proceeding with the administration of the study vaccine.
* Lymphoproliferative disorder or malignancy within 5 years before study vaccination (excluding effectively treated non-melanoma skin cancer).

Prior/Concomitant therapy

* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study intervention(s) during the period beginning 30 days before the first doses (Day -29 to Day 1), or their planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol within the period starting 30 days before the first dose and ending 30 days after the last dose of study intervention(s)* administration with the exception of any licensed influenza vaccine which may be administered ≥ 15 days before or after study vaccinations (dTpa and RSV maternal vaccines).

  * *In case emergency mass vaccination for an unforeseen public health threat (e.g. a pandemic) is organized by public health authorities outside the routine immunization program, the time period described above can be reduced if necessary for that vaccine (if it is used according to the local governmental recommendations and that the Sponsor is notified accordingly). Therefore, COVID-19 vaccines will be allowed, when administered ≥ 15 days before or after study vaccinations (dTpa and RSV maternal vaccines).
* Administration of long-acting immune-modifying drugs at any time during the study period (e.g. infliximab).
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before the administration of the first dose of study intervention(s) or planned administration during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first study intervention dose(s) to 2 months after first vaccination. For corticosteroids, this will mean prednisone equivalent ≥5 mg/day for adult participants/ ≥0.5 mg/kg/day. Inhaled and topical steroids are allowed.
* Previous experimental vaccination against RSV.
* Boostrix (dTpa) administration for which the vaccination is not aligned with the local recommendations for dTap vaccination or not aligned with the locally approved Boostrix (dTpa) prescribing information.

Prior/Concurrent clinical study experience

• Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational intervention (drug/invasive medical device).

Other exclusions

* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Alcoholism or substance use disorder within the past 24 months based on the presence of two or more of the following abuse criteria: hazardous use, social/interpersonal problems related to use, neglected major roles to use, withdrawal tolerance, use of larger amounts or longer, repeated attempts to quit or control use, much time spent using, physical or psychological problems related to use, activities given up to use, craving.
* Any study personnel or their immediate dependents, family, or household members.
* Child in care.

Ages: 9 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Beaumont, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned to enroll 252 participants in 4 groups as per Protocol. However, due to early stoppage of enrolment and further vaccination, only 9 participants were enrolled in the study, out of which 8 participants were assigned to individual groups, except for the dTpa_RSV-P group, hence this group was not included in the results record.
Pre-assignment Details: Out of the 9 participants enrolled in the study, 1 participant withdrew consent before being assigned to any of the groups and was not vaccinated. 8 participants were vaccinated and were included in the Exposed set.
Period: Overall Study
Arm/Group | RSV_dTpa-P Group | RSV_dTpa-A Group | dTpa_RSV-A Group
Started | 1 | 3 | 4
Completed | 1 | 3 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV_dTpa-P Group | RSV_dTpa-A Group | dTpa_RSV-A Group | Total
Number analyzed (Participants) | 1 | 3 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age and its descriptive analysis is presented for adult participants only. There was only one participant in the pediatric age group, hence the mean and standard deviation could not be calculated. Since the actual age is considered personal information (PI) attributable to the participant and it will increase the risk of re-identification, it will not be disclosed in the record.
  Years | NA (NA) — There was only one participant in the pediatric age group, hence the mean and standard deviation could not be calculated. Since the actual age is considered personal information (PI) attributable to the participant and it will increase the risk of re-identification, it will not be disclosed in the record. | 42.3 (2.5) | 38.0 (9.4) | 39.9 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 8
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  BLACK OR AFRICAN AMERICAN | 1 | 0 | 0 | 1
  WHITE | 0 | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Any Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or results in abnormal pregnancy outcomes. Any is defined as the occurrence of the symptom regardless of intensity grade or relationship to vaccination.
Time Frame: During the entire study period (from Day 1 up to Day 181)
Population: The analysis was performed on the Exposed Set, which included all participants who received the study intervention (RSV maternal vaccine or dTpa vaccine).
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_dTpa-P Group | RSV_dTpa-A Group | dTpa_RSV-A Group
Number analyzed (Participants) | 1 | 3 | 4
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Adverse Events (AEs)/SAEs Leading to Study Withdrawal
Description: An AE is any untoward medical occurrence, symptom, or disease in a clinical study participant that is temporally associated with the study intervention. The AE may or may not be considered related to the study intervention.
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or results in abnormal pregnancy outcomes.
  A participant is considered to have withdrawn from the study if no new study procedure has been performed or no new information has been collected for him/her since the date of withdrawal/last contact.
Time Frame: During the entire study period (from Day 1 up to Day 181)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_dTpa-P Group | RSV_dTpa-A Group | dTpa_RSV-A Group
Number analyzed (Participants) | 1 | 3 | 4
Participants | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Any Solicited Administration Site Events
Description: Assessed solicited administration site events include pain, erythema and swelling. Any pain = occurrence of the symptom regardless of intensity grade. Any erythema and swelling = symptom reported with a surface diameter lower than or equal to 20 millimeters.
Time Frame: During the 7 days follow-up period post-Dose 1
Population: The analysis was performed on the Solicited Safety Set, which included all participants in the Exposed Set who have solicited safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_dTpa-P Group | RSV_dTpa-A Group | dTpa_RSV-A Group
Number analyzed (Participants) | 1 | 3 | 4
Participants
  Pain | 1 | 1 | 3
  Erythema | 0 | 0 | 1
  Swelling | 0 | 0 | 0

4. Primary Outcome: Number of Participants Reporting Any Solicited Systemic Events
Description: Assessed solicited systemic events include fatigue, headache, gastrointestinal (GI) symptoms (nausea, vomiting, diarrhea, abdominal pain) and fever. The preferred location for measuring temperature is the oral cavity. Fever is defined as temperature equal to or above (≥) 38.0 °C/100.4°F. Any is defined as the occurrence of the symptom regardless of intensity grade.
Time Frame: During the 7 days follow-up period post-Dose 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_dTpa-P Group | RSV_dTpa-A Group | dTpa_RSV-A Group
Number analyzed (Participants) | 1 | 3 | 4
Participants
  Fatigue | 0 | 1 | 1
  Headache | 0 | 1 | 2
  Nausea | 0 | 1 | 0
  Vomiting | 0 | 0 | 0
  Diarrhea | 0 | 2 | 2
  Abdominal pain | 0 | 1 | 0
  Fever | 0 | 0 | 0

5. Primary Outcome: Number of Participants Reporting Any Unsolicited AEs
Description: An unsolicited AE is an event reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event. Any is defined as the occurrence of the unsolicited AE regardless of intensity grade or relationship to vaccination.
Time Frame: During the 30 days follow-up period post-Dose 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_dTpa-P Group | RSV_dTpa-A Group | dTpa_RSV-A Group
Number analyzed (Participants) | 1 | 3 | 4
Participants | 0 | 1 | 1

6. Primary Outcome: Number of Participants Reporting SAEs and Medically Attended Adverse Events (MAEs)
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or results in abnormal pregnancy outcomes.
  An MAE is an unsolicited AE for which the participants receive medical attention, defined as symptoms or illnesses requiring a hospitalization, or an emergency room visit, or visit to/by a health care provider.
Time Frame: During the 30 days follow-up period post-Dose 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_dTpa-P Group | RSV_dTpa-A Group | dTpa_RSV-A Group
Number analyzed (Participants) | 1 | 3 | 4
Participants | 0 | 0 | 0

7. Primary Outcome: Number of Participants Reporting AEs/SAEs/MAEs Leading to Study Withdrawal
Description: An AE is any untoward medical occurrence, symptom, or disease in a clinical study participant that is temporally associated with the study intervention. The AE may or may not be considered related to the study intervention.
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or results in abnormal pregnancy outcomes.
  An MAE is an unsolicited AE for which the participants received medical attention defined as symptoms or illnesses requiring a hospitalization, or an emergency room visit, or visit to/by a health care provider.
  A participant is considered to have withdrawn from the study if no new study procedure has been performed or no new information has been collected for him/her since the date of withdrawal/last contact.
Time Frame: During the 30 days follow-up period post-Dose 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RSV_dTpa-P Group | RSV_dTpa-A Group | dTpa_RSV-A Group
Number analyzed (Participants) | 1 | 3 | 4
Participants | 0 | 0 | 0

8. Secondary Outcome: RSV-A Neutralizing Antibody Titers for Participants in RSV_dTpa-P Group and RSV_dTpa-A Group at Day 1
Description: RSV-A neutralizing antibody titer expressed in Estimated Dose: serum dilution giving a 60% reduction of the signal compared to a control without serum (ED60) is presented for each participant who received the RSV MAT vaccine and was assigned to the respective group.
Time Frame: At pre-dosing (Day 1)
Population: Due to a small number of participants assigned to the study groups, geometric mean titers could not be summarized for this outcome measure. Hence, antibody titer was reported for each participant evaluated in the respective arm, who received the RSV MAT vaccine and had individual immunogenicity data available at the specified time point.
Measure: Number; unit: Titers (ED60)
Arm/Group | RSV_dTpa-P Group | RSV_dTpa-A Group
Number analyzed (Participants) | 1 | 3
Titers (ED60)
  Participant 1: number analyzed (Participants) | 1 | 1
  Participant 1 | 86 | 1355
  Participant 2: number analyzed (Participants) | 0 | 1
  Participant 2 |  | 792
  Participant 3: number analyzed (Participants) | 0 | 1
  Participant 3 |  | 177

9. Secondary Outcome: RSV-A Neutralizing Antibody Titers for Participants in RSV_dTpa-P Group and RSV_dTpa-A Group at Day 31
Description: RSV-A neutralizing antibody titer expressed in ED60 is presented for each participant who received the RSV MAT vaccine and was assigned to the respective group.
Time Frame: At 30 days post-RSV MAT vaccine administration (Day 31)
Population: as for outcome 8
Measure: Number; unit: Titers (ED60)
Arm/Group | RSV_dTpa-P Group | RSV_dTpa-A Group
Number analyzed (Participants) | 1 | 3
Titers (ED60)
  Participant 1: number analyzed (Participants) | 1 | 1
  Participant 1 | 1702 | 21707
  Participant 2: number analyzed (Participants) | 0 | 1
  Participant 2 |  | 38258
  Participant 3: number analyzed (Participants) | 0 | 1
  Participant 3 |  | 17765

10. Secondary Outcome: RSV-B Neutralizing Antibody Titers for Participants in RSV_dTpa-P Group and RSV_dTpa-A Group at Day 1
Description: RSV-B neutralizing antibody titer expressed in ED60 is presented for each participant who received the RSV MAT vaccine and was assigned to the respective group.
Time Frame: At pre-dosing (Day 1)
Population: as for outcome 8
Measure: Number; unit: Titers (ED60)
Arm/Group | RSV_dTpa-P Group | RSV_dTpa-A Group
Number analyzed (Participants) | 1 | 3
Titers (ED60)
  Participant 1: number analyzed (Participants) | 1 | 1
  Participant 1 | 373 | 2434
  Participant 2: number analyzed (Participants) | 0 | 1
  Participant 2 |  | 525
  Participant 3: number analyzed (Participants) | 0 | 1
  Participant 3 |  | 461

11. Secondary Outcome: RSV-B Neutralizing Antibody Titers for Participants in RSV_dTpa-P Group and RSV_dTpa-A Group at Day 31
Description: as for outcome 10
Time Frame: At 30 days post-RSV MAT vaccine administration (Day 31)
Population: as for outcome 8
Measure: Number; unit: Titers (ED60)
Arm/Group | RSV_dTpa-P Group | RSV_dTpa-A Group
Number analyzed (Participants) | 1 | 3
Titers (ED60)
  Participant 1: number analyzed (Participants) | 1 | 1
  Participant 1 | 2089 | 138336
  Participant 2: number analyzed (Participants) | 0 | 1
  Participant 2 |  | 14233
  Participant 3: number analyzed (Participants) | 0 | 1
  Participant 3 |  | 34743

12. Secondary Outcome: RSV MAT Immunoglobulin G (IgG) Antibody Concentrations for Participants in RSV_dTpa-P Group and RSV_dTpa-A Group at Day 1
Description: RSV MAT IgG antibody concentration expressed in ELISA units per milliliter (EU/mL) is presented for each participant who received the RSV MAT vaccine and was assigned to the respective group.
Time Frame: At pre-dosing (Day 1)
Population: Due to a small number of participants assigned to the study groups, geometric mean concentrations could not be summarized for this outcome measure. Hence, antibody concentration was reported for each participant evaluated in the respective arm, who received the RSV MAT vaccine and had individual immunogenicity data available at the specified time point.
Measure: Number; unit: EU/mL
Arm/Group | RSV_dTpa-P Group | RSV_dTpa-A Group
Number analyzed (Participants) | 1 | 3
EU/mL
  Participant 1: number analyzed (Participants) | 1 | 1
  Participant 1 | 1949 | 4967
  Participant 2: number analyzed (Participants) | 0 | 1
  Participant 2 |  | 3279
  Participant 3: number analyzed (Participants) | 0 | 1
  Participant 3 |  | 4727

13. Secondary Outcome: RSV MAT IgG Antibody Concentrations for Participants in RSV_dTpa-P Group and RSV_dTpa-A Group at Day 31
Description: RSV MAT IgG antibody concentration expressed in EU/mL is presented for each participant who received the RSV MAT vaccine and was assigned to the respective group.
Time Frame: At 30 days post-RSV MAT vaccine administration (Day 31)
Population: as for outcome 12
Measure: Number; unit: EU/mL
Arm/Group | RSV_dTpa-P Group | RSV_dTpa-A Group
Number analyzed (Participants) | 1 | 3
EU/mL
  Participant 1: number analyzed (Participants) | 1 | 1
  Participant 1 | 50193 | 149510
  Participant 2: number analyzed (Participants) | 0 | 1
  Participant 2 |  | 218190
  Participant 3: number analyzed (Participants) | 0 | 1
  Participant 3 |  | 402812

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected during the 7-day follow-up period after vaccination. Unsolicited AEs were collected during the 30-day follow-up period after vaccination. SAEs were collected from study start (Day 1) up to 180 days after vaccination (Day 181).
Arm/Group | RSV_dTpa-P Group | RSV_dTpa-A Group | dTpa_RSV-A Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 1/1 | 2/3 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV_dTpa-P Group (N=1) | RSV_dTpa-A Group (N=3) | dTpa_RSV-A Group (N=4)
Administration site pain (General disorders) | 1 (1) | 1 (1) | 3 (9)
Fatigue (General disorders) | 0 (0) | 1 (5) | 1 (2)
Administration site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (3) | 2 (2)
Hypomenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT05169905/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/05/NCT05169905/SAP_001.pdf